CLINICAL TRIAL: NCT00830232
Title: Effects of Carotid Stent Design on Cerebral Embolization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carlos H. Timaran, Vascular and Endovascular Surgeon, Dallas VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB#08-035
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Stroke; Carotid Stenosis
Keywords: Stroke; Carotid stenosis; stents
MeSH Terms: conditions — Stroke; Carotid Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed-cell stent (Xact stent) (Active Comparator): For patients randomized to the closed-cell stent group, the Xact closed-cell stents were used. The Xact stent is a FDA approved device.
  Interventions: Device: closed-cell stent (Xact stent)
- Open-cell stent (Acculink carotid) (Active Comparator): For patients randomized to the open-cell stent group, the Acculink carotid stent was used. The Acculink stent is a FDA approved device.
  Interventions: Device: Open-cell stent (Acculink carotid)

INTERVENTIONS:
Device: closed-cell stent (Xact stent) — Patients enrolled in this study arm underwent for carotid stenting using closed stent cell. The graft used in this groups was the Xact closed-cell stent. This type of device is rigid device with dense conposition of the nitinol rigns.
  Carotid stenting was used on standard fashion using filters as embolic protection device.
  Other Names: Carotid artery angioplasty
  Arms: Closed-cell stent (Xact stent)
Device: Open-cell stent (Acculink carotid) — Patients enrolled in this study arm underwent for carotid stenting using open stent cell stents. This type of stent is a tube shaped graft composed of flexible nitinol rings. The device used in this group was the Acculinx open-cell stent.
  Stenting procedure eas performed on standard fashion.Filters were used as embolic protection device.
  Other Names: Carotid artery angioplasty
  Arms: Open-cell stent (Acculink carotid)

SUMMARY:
The goal of the proposed study is to contrast the relative efficacy of closed-cell stents versus open-cell stents in preventing periprocedural cerebral embolization in high-risk patients with symptomatic and asymptomatic extracranial carotid stenosis undergoing carotid artery stenting (CAS).

DETAILED DESCRIPTION:
Stroke is responsible for more than 10% of all deaths and much severe disability in developed countries. In the United States, approximately 600,000 new strokes are reported annually, of which 150,000 are fatal, and more than 4,000,000 surviving stroke victims are affected by significant disability. Seventy-five percent of strokes occur in the distribution of the carotid arteries and are considered of a thromboembolic etiology, most of which originate in carotid lesions. Carotid artery stenting (CAS) with cerebral embolic protection is currently the preferred treatment of carotid stenosis in high risk surgical patients, i.e., those with significant comorbidities or a hostile neck from previous surgical procedures or radiation. Although several predictors of adverse outcomes after CAS have been identified, the effects of device characteristics, including stent design, on neurologic adverse events have not been established.

The proposed study will be a randomized prospective controlled trial designed to test the hypothesis that the implantation of closed-cell stents for carotid lesions in high-risk patients will be associated with a reduced perioperative cerebral microembolization, as detected by transcranial Doppler and diffusion-weighted magnetic resonance imaging of the brain, and reduced 30-day stroke, myocardial infarction, and death rates when compared with the implantation of open-cell stents.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at high risk for carotid endarterectomy due to either anatomic or co-morbid conditions; AND
* Symptomatic patients (TIA or non-disabling stroke within 6 months of the procedure), with carotid stenosis ≥ 50% as diagnosed by angiography, using NASCET methodology (50); OR
* Asymptomatic patients with carotid stenosis ≥ 80% as diagnosed by angiography, using NASCET methodology

Exclusion Criteria:

* Conditions that interfere with the evaluation of endpoints
* Subject has anticipated or potential sources of cardiac emboli
* Subject plans to have a major surgical procedure within 30 days after the index procedure.
* Subject has intracranial pathology that makes the subject inappropriate for study participation.
* Subject has a total occlusion of the ipsilateral carotid artery (i.e., CCA).
* Severe circumferential lesion calcification that may restrict the full deployment of the carotid stent.
* Carotid stenosis located distal to the target stenosis that is more severe than the target stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos H Timaran, MD, Principal Investigator — Dallas VA Medical Center
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Timaran CH, Rosero EB, Higuera A, Ilarraza A, Modrall JG, Clagett GP. Randomized clinical trial of open-cell vs closed-cell stents for carotid stenting and effects of stent design on cerebral embolization. J Vasc Surg. 2011 Nov;54(5):1310-1316.e1; discussion 1316. doi: 10.1016/j.jvs.2011.05.013. Epub 2011 Jul 1. PMID 21723064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruitment was started on december 2008 and continued until February 2012. Patients recruitment and consenting were performed at the medical clinic.
Pre-assignment Details: Patients were considered officially enrolled after the randomization, which was performed during the procedure after the initial angiography (initial image of the brain blood flow).
Groups:
- Closed-cell Stent: Patients enrolled in this study arm underwent for carotid stenting using closed stent cell. The graft used in this group was the Xact closed-cell stent. This type of device is a rigid device with a dense composition between the nitinol rings.
  Carotid stenting was used on standard fashion using filters as embolic protection device.
- Open-cell Stent: Patients enrolled in this study arm underwent for carotid stenting using open stent cell stents. This type of stent is a tube shaped graft composed of flexible nitinol rings. The device used in this group was the Acculinx open-cell stent.
  Stenting procedure eas performed on standard fashion.Filters were used as embolic protection device.
Period: Overall Study
Arm/Group | Closed-cell Stent | Open-cell Stent
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Closed-cell Stent: closed-cell stent : Closed-cell stent: Comparison of two types of carotid stent designs (open- vs. closed-cell) regarding the primary and secondary outcomes.
- Open-cell Stent: Open-cell stent : Open-cell Stent: Comparison of two types of carotid stent designs (open- vs. closed-cell) regarding the primary and secondary outcomes.
- Total: Total of all reporting groups
Arm/Group | Closed-cell Stent | Open-cell Stent | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8.07) | 67 (8.5) | 66.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 17 | 19 | 36
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Transcranial Doppler Counts of Micro-embolic Signals in the Ipsilateral Middle Cerebral Artery.
Description: Bilateral transcranial Doppler scan monitoring of the anterior and middle cerebral arteries was performed using a PMD150-ST3 digital transcranial Doppler pulsed-wave ultrasound scan system (Spencer Technologies, Seattle, Wash) with 2-MHz probes located over the temporal bones above the zygomatic arch. Isolated microembolic signals (MES) were identified from Doppler spectras according to the criteria given by the Consensus Committee of the Ninth International Cerebral Hemodynamic Symposium. If the number of MES was too high to be counted separately, heartbeats with microemboli were counted as microembolic showers. To avoid confusion, MES detected during contrast injection were excluded from the analysis. For analysis purposes, the procedure was divided into the following phases: lesion crossing, filter deployment, IVUS examination, predilation, stent deployment, postdilatation (when applicable), and filter removal.
Time Frame: First 24 hours after implantation of carotid stent
Measure: Median (Inter-Quartile Range); unit: Micro-emboli
Arm/Group | Closed-cell Stent | Open-cell Stent
Number analyzed (Participants) | 20 | 20
Micro-emboli | 264 [222 to 343] | 339 [163 to 408]

2. Secondary Outcome: Composite of Any Stroke, Myocardial Infarction or Death
Time Frame: within 30 days after the carotid stenting procedure
Reporting Status: Not Posted

3. Secondary Outcome: Subclinical Cerebral Embolization Assessed by Brain Diffusion-weighted MRI
Time Frame: within 24 hours after carotid artery stenting
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessment for adverse events was perfumed at 30 days after carotid stenting.
Description: Only serious adverse events were collected/assessed for this study
Arm/Group | Closed-cell Stent | Open-cell Stent
Serious Adverse Events (participants affected / at risk) | 7/20 | 4/20
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed-cell Stent (N=20) | Open-cell Stent (N=20)
Non-ST elevation myocardial infarction (NSTEMI) (Cardiac disorders) | 2 (2) | 0 (0)
Groin Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Peri-operative hypotension (Vascular disorders) | 3 (3) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Angina (Cardiac disorders) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Transient Ischemic Atack (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
1. Small sample size 2.randomization did not eliminate all pretreatment differences between groups because of the small sample size.3.All patients underwent Stenting under ﬁlter embolic protection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No